CLINICAL TRIAL: NCT05629247
Title: Pediatric Intensive Care Unit and Primary Immune Deficiency
Acronym: PICUPID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17-158
Record Dates: First submitted 2018-06-12; First posted 2022-11-29 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Immuno-Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Screening (Other)
  Interventions: Diagnostic Test: Systematic screening of immune deficiency

INTERVENTIONS:
Diagnostic Test: Systematic screening of immune deficiency — Systematic screening of immune deficiency with blood tests

SUMMARY:
To date, many studies have focused on the characteristics of PID in children, allowing to highlight an entry into the disease in the context of more or less severe infections in all pediatric departments. However, only one study has so far studied the frequency of these PID in a pediatric resuscitation unit, which is why we propose this study to the Caen University Hospital.

Investigtors propose a two-step study, both retrospective and prospective, in order to increase our cohort.

The retrospective analysis of the data will be done over the period 2013-2016, the prospective analysis will be done from May 2017 to January 2018. The study will be monocentric, performed in the pediatric resuscitation department of the University Hospital of Caen to evaluate the prevalence of PIDs and describe their characteristics.

The included patients will be aged 0 to 18 years, hospitalized in the pediatric intensive care unit for a serious infection and / or of an unfavorable evolution, or an opportunistic germ infection in the absence of a DIP or an immunodeficiency previously known. The inclusion will be proposed by the intensive care pediatricians. Authorization by the legal representative will be required in advance.

The data will be collected during the systematic consultation in pediatric haemato-immuno-oncology within 3 months after their hospitalization in intensive care unit to detect a DIP by a thorough interrogation, a clinical examination and a first-line biological assessment.

A second consultation will be scheduled in the 3 months following the 1st with announcement of the results of the first balance sheet and completion of a second complementary balance sheet if a suspicion of DIP persists at the end of the first balance sheet.

The precise description of the incidence of these immunodeficiencies and their characteristics could lead to the development of recommendations on the routine screening of PID in pediatric resuscitation; an early diagnosis enabling preventive and curative management (vaccine, immunoglobulin, antibiotic prophylaxis, etc.) to be put in place in order to limit the risk of infectious recurrence and reduce the morbidity.

ELIGIBILITY:
Inclusion Criteria:

Any child hospitalized in the Pediatric Resuscitation Unit for:

* Severe sepsis or septic shock including those without microbiological documentation or portal of entry found.
* ≥ 1 documented invasive infection with encapsulated germ (Streptococcus pneumoniae, group A streptococcus, Haemophilus influenzae, Neisseria meningitidis).
* An invasive infection with an unusual germ or an opportunistic infection: Bacterial: Salmonella, Tuberculosis, / Fungal: Aspergillosis, Cryptococcosis, Candidiasis / Parasitic: Toxoplasmosis, Pneumocystosis, Giarda lamblia / Viral: enterovirus, CMV, EBV, viral encephalitis

Exclusion Criteria:

* Patient with known primary or secondary immunodeficiency: HIV, known neoplasia, immunosuppressive or immunomodulatory therapy, renal failure, nephrotic syndrome, hypoprotidemia, cirrhosis with hepatic insufficiency, sickle cell disease, splenectomy.
* Local-regional factors that may be responsible for infections: foreign body in the airways, history of ENT surgery or neurosurgery, history of fracture of the skull base, cystic fibrosis, chronic respiratory insufficiency.
* Refusal to sign the consent of the legal representative.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Actual)
Dates: Start 2018-01-26 (Actual); Primary Completion 2019-01-26 (Actual); Study Completion 2020-01-26 (Actual)

PRIMARY OUTCOMES:
primary immunodeficiencies | change between baseline and 3 month after baseline
  to detect primary immunodeficiencies in the course of serious infections or of unfavorable evolution in patients requiring care in the pediatric resuscitation department

CONTACTS AND LOCATIONS:
Locations (1):
- Caen University Hospital, Caen, France

IPD SHARING:
Plan to Share IPD: No